CLINICAL TRIAL: NCT04074265
Title: Efficacy of a Peri-Operative Surgical-Site, Multimodal Drug Injection in Pediatric Patients With Cerebral Palsy Undergoing Hip Surgery: A Randomized Controlled Trial
Brief Title: Peri-operative Use of a Pain Injection in Pediatric Patients With Cerebral Palsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Rachel Thompson, MD, Associate Director, Center for Cerebral Palsy, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-001423
Record Dates: First submitted 2019-08-27; First posted 2019-08-30 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy; Hip Dysplasia; Pain, Postoperative
Keywords: cerebral palsy; randomized controlled trial; pediatric; pain management; perioperative medicine
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation; Pain, Postoperative; Agnosia | interventions — Ropivacaine; Ketorolac; Epinephrine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to either treatment/intervention group or placebo. All other aspects of care will be identical between the two groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Surgeon, participant, and all nursing staff involved in recording post-operative outcomes will be blinded to treatment group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain injection (Active Comparator): This group will be injected with a cocktail totaling 40mL (20mL on each side) that will be composed of ropivicaine 2mg/mL (3mg/kg), epinephrine 1mg/mL (0.5mg), ketorolac 30mg/mL (0.5mg/kg).
  Interventions: Drug: Ropivacaine injection
- Normal saline (Placebo Comparator): The control group will receive an injection of 40mL of 0.9% sodium chloride solution.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Ropivacaine injection — Injection containing a mix of the above medications will be performed while the patient is still under general anesthesia, following wound closure, and will be injected evenly between the deep and superficial tissues in an extra-articular pattern (no injection of the synovium or capsule).
  Other Names: ropivacaine; ketorolac; epinephrine
  Arms: Pain injection
Drug: normal saline — Injection containing normal saline will be performed while the patient is still under general anesthesia, following wound closure, and will be injected evenly between the deep and superficial tissues in an extra-articular pattern (no injection of the synovium or capsule).
  Arms: Normal saline

SUMMARY:
Pain management in pediatric patients presents a difficult challenge. Unlike adults, pediatric patients often cannot communicate their pain management needs clearly. Adequate pain control after surgery is pivotal for these patients in order to prevent negative physiologic and psychologic complications and to improve surgical outcomes. There is an ongoing shift away from the use of opioids in the post-operative setting due to both their negative side effects and their high potential for dependence and abuse.

A variety of new techniques of multimodal pain management have been developed and utilized in elective orthopaedic procedures. Injection of local anesthetics is becoming a widely popular technique utilized in adult arthroplasty. This technique blocks pain directly at the site of injection, and therefore can improve post-operative pain while minimizing side effects. Evidence has demonstrated this technique to be both safe and effective, resulting in reduced opioid consumption post-operatively. However, this technique has not been studied for use in pediatric patients, a population in which reduced narcotic use is equally, if not more important than in adult patients.

This study is a prospective, randomized controlled trial with 2 parallel arms. The goal of this study is to assess the efficacy of a surgical-site pain injection administered in pediatric patients with cerebral palsy undergoing major hip surgery. Patients who are scheduled to undergo surgery will be randomized to either intervention (injection of a pain cocktail) or placebo (injection of normal saline). The pain cocktail includes three medications: ropivacaine (a local anesthetic), ketorolac (an anti-inflammatory medication), and epinephrine (a medication to constrict blood vessels and increase the duration of action of any co-administered medications). A surgeon who is blinded to treatment group will administer the injection at the end of the procedure, prior to the patient waking from anesthesia. The injection is in addition to our typical multi-modal pain control protocol, which includes epidural anesthesia, acetaminophen, anti-inflammatories, oral narcotics and anti-spasmodic agents. Patients will then be monitored post-operatively and pain medication consumption (both while in the hospital post-operatively and for the first two weeks following discharge), patient-reported and/or nurse-recorded pain scores, length of hospital stay, and adverse effects will be recorded. At the first post-operative visit, patients' parents will be asked to complete a survey designed to assess parent satisfaction with their child's pain management after surgery. Patients, parents, and surgeons will be blinded to treatment group allocation. Data will be collected while the patient is in the hospital, after surgery (average duration 3-4 days), and at the first post-operative visit two to three weeks after surgery.

DETAILED DESCRIPTION:
With the ongoing opioid epidemic in the United States, there has been a shift toward the use of non-opioid alternatives for pain control in the post-operative period. The development of a multimodal approach to pain management has seen a rise in the use of local anesthesia, whether as a peripheral nerve block or as an peri/intra-articular injection. These techniques have shown to be very effective in the adult population for improving pain and reducing the need for opioid consumption post-operatively. However, these techniques have yet to be studied in the pediatric population. The purpose of this study is to examine the efficacy of a local anesthetic injection post-operatively in pediatric patients with cerebral palsy undergoing major surgery as part of a multi-modal pain control protocol. The investigators hypothesize that peri-articular injection of a pain cocktail containing a mix of local anesthetic, anti-inflammatory medication, and epinephrine at the end of surgery will result in decreased opioid use in the immediate peri-operative period in pediatric patients with cerebral palsy undergoing proximal femoral osteotomy when compared to an injection of normal saline. The investigators also hypothesize that the pain injection will result in decreased mean pain scores post-operatively, shorter hospital stays and improved parent satisfaction when compared to normal saline injection. With this study, the investigators hope to provide evidence to support the use of a minimally invasive, safe-to-use pain injection that will reduce the need for opioids in pediatric patients undergoing orthopaedic procedures.

Study Design:

This study is a prospective, randomized controlled trial with 2 parallel arms. Patients will be randomly assigned to the 2 treatment groups: surgical-site injection with ropivacaine, ketorolac, and epinephrine, or surgical-site injection with normal saline. Randomization will be performed via random number generator and will be carried out by a research associate who will not participate in study recruitment or outcomes assessment. Allocations will be concealed on a password-protected database accessible only to the research associate. Patients, surgeons, and nursing staff who perform post-operative assessments will be blinded to treatment allocation.

Surgical Procedure:

Patients undergoing unilateral or bilateral hip proximal femoral osteotomies will be included in the study. All patients will be treated with standard-of-care techniques chosen by the treating surgeon. The addition of pelvic osteotomies and/or soft tissue procedures will be at the discretion of the treating surgeon and will not exclude the patient from the study. Written consent will be obtained for all patients prior to the surgical procedure. Parental consent will be obtained, in addition to patient assent for all patients of appropriate age and intellectual capability. All patients will have a general anesthetic with a lumbar epidural. No preemptive scheduled analgesic regimen will be employed. All medications administered during induction and maintenance of anesthesia will be managed by the anesthesiologist and titrated at their discretion.

The local anesthetic group will be injected with a cocktail totaling 40 milliliters (mL) (20mL on each side) that will be composed of ropivicaine 2mg/mL (3mg/kg), epinephrine 1mg/mL (0.5mg), ketorolac 30mg/mL (0.5mg/kg). The control group will receive 40mL of 0.9% sodium chloride solution. The injection will be performed while the patient is still under general anesthesia, following wound closure, and will be injected evenly between the deep and superficial tissues in an extra-articular pattern (no injection of the synovium or capsule). All injections will be performed using a 20-gauge needle. All medications will be obtained from the hospital pharmacy. All injections will be prepared by an operating room nurse under the supervision of a research assistant, and placed in an unlabeled syringe to allow for blinding of the surgeon administering the injection.

Post-Operative Protocol:

The epidural anesthesia will be started at the discretion of the attending anesthesiologist either before or on-arrival to the post-anesthesia care unit. Any additional medications administered during the immediate post-operative period in the post-anesthesia care unit will be prescribed by the attending anesthesiologist and will not be standardized. Beginning when the patient leaves the post-anesthesia care unit, all patients will be given the following pain regimen: acetaminophen (15mg/kg PO or per g-tube every 6 hours around the clock), ketorolac (0.5mg/kg IV every 8 hours for 3 doses) followed by ibuprofen (10mg/kg PO or per g-tube every 8 hours as needed for mild pain (pain score 1-3)), diazepam (0.1mg/kg PO or per g-tube every 6 hours around the clock for 36 hours followed by every 6 hours as needed for muscle spasms), and oxycodone (0.1mg/kg PO or per g-tube every 6 hours as needed for severe pain (pain score 7-10)). Nurses will be instructed to offer this as-needed medication to patients at standardized intervals every 4 hours when performing pain assessments. Additional medication for pain may be administered if the protocol does not result in adequate pain relief, at the discretion of the treating physician. The epidural will be titrated by the acute pain anesthesiology team for inadequate pain control, and all epidurals will be discontinued the morning of post-operative day two. All patients will be discharged on a standardized medication regimen as follows: diazepam (0.1mg/kg PO or per g-tube every 6 hours for 14 days), oxycodone (0.5mg/kg PO or per g-tube every 6 hours as needed for severe pain, 20 doses), acetaminophen (15mg/kg PO or per g-tube every 6 hours for 14 days), and ibuprofen (10mg/kg PO or per g-tube every 8 hours for 14 days). Inpatient and outpatient narcotic consumption will be recorded as morphine equivalents per kilogram, to allow adjustment for the weight-based dosing used in pediatric patients.

All other aspects of post-operative care, including (but not limited to) physical therapy, weight bearing status, mobilization, and bracing will be decided on a case-by-case basis by the treating surgeon.

Data Collection and Protection:

Data will be collected by approved research personnel via access to the medical record. Personal identifying information collected will include name, date of birth, medical record number, and telephone number. All data will be labeled with a code that can be linked to this personal identifying information. Data will be collected only from the hospitalization following the surgical procedure and from the first post-operative visit. This data will include: narcotic consumption, pain scores, complications or adverse events, and re-admission in the immediate post-operative period (first two weeks post-operatively). All data will be stored on a secure, encrypted data storage device or password protected and encrypted internet-based storage device.

ELIGIBILITY:
Inclusion Criteria:

* under 18 years old
* diagnosis of cerebral palsy
* undergoing uni- or bilateral proximal femoral osteotomy

Exclusion Criteria:

* ongoing preoperative opioid use
* history of allergic reaction to any component of the pain injection

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M Thompson, MD, Principal Investigator — University of California, Los Angeles
Locations (4):
- United States (4):
  - Orthopaedic Institute for Children, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen JD, Casavant MJ, Spiller HA, Chounthirath T, Hodges NL, Smith GA. Prescription Opioid Exposures Among Children and Adolescents in the United States: 2000-2015. Pediatrics. 2017 Apr;139(4):e20163382. doi: 10.1542/peds.2016-3382. Epub 2017 Mar 20. PMID 28320869
- [Background] Andersen KV, Pfeiffer-Jensen M, Haraldsted V, Soballe K. Reduced hospital stay and narcotic consumption, and improved mobilization with local and intraarticular infiltration after hip arthroplasty: a randomized clinical trial of an intraarticular technique versus epidural infusion in 80 patients. Acta Orthop. 2007 Apr;78(2):180-6. doi: 10.1080/17453670710013654. PMID 17464604
- [Background] Chaw S, Lo Y, Shariffuddin II, Wong J, Lee J, Leong DW, Ng KW, Chan L. Evaluation of the quality of acute pain management in a pediatric surgical setting: Validation of a parent proxy modified version of the revised American Pain Society Patient Outcome Questionnaire. Paediatr Anaesth. 2019 Jan;29(1):68-76. doi: 10.1111/pan.13528. Epub 2018 Oct 31. PMID 30381868
- [Background] Harbaugh CM, Lee JS, Hu HM, McCabe SE, Voepel-Lewis T, Englesbe MJ, Brummett CM, Waljee JF. Persistent Opioid Use Among Pediatric Patients After Surgery. Pediatrics. 2018 Jan;141(1):e20172439. doi: 10.1542/peds.2017-2439. Epub 2017 Dec 4. PMID 29203521
- [Background] Koehler D, Marsh JL, Karam M, Fruehling C, Willey M. Efficacy of Surgical-Site, Multimodal Drug Injection Following Operative Management of Femoral Fractures: A Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Mar 15;99(6):512-519. doi: 10.2106/JBJS.16.00733. PMID 28291185
- [Background] Nolan J, Chalkiadis GA, Low J, Olesch CA, Brown TC. Anaesthesia and pain management in cerebral palsy. Anaesthesia. 2000 Jan;55(1):32-41. doi: 10.1046/j.1365-2044.2000.01065.x. PMID 10594431
- [Background] Troelsen A, Elmengaard B, Soballe K. A new minimally invasive transsartorial approach for periacetabular osteotomy. J Bone Joint Surg Am. 2008 Mar;90(3):493-8. doi: 10.2106/JBJS.F.01399. PMID 18310698
- [Background] Vendittoli PA, Makinen P, Drolet P, Lavigne M, Fallaha M, Guertin MC, Varin F. A multimodal analgesia protocol for total knee arthroplasty. A randomized, controlled study. J Bone Joint Surg Am. 2006 Feb;88(2):282-9. doi: 10.2106/JBJS.E.00173. PMID 16452738

RESULTS

PARTICIPANT FLOW:
Groups:
- Pain Injection: This group will be injected with a cocktail totaling 50mL (25mL on each side) that will be composed of ropivicaine 2mg/mL (3mg/kg), epinephrine 1mg/mL (0.5mg), ketorolac 30mg/mL (0.5mg/kg).
  Ropivacaine injection: Injection containing a mix of the above medications will be performed while the patient is still under general anesthesia, following wound closure, and will be injected evenly between the deep and superficial tissues in an extra-articular pattern (no injection of the synovium or capsule).
- Normal Saline: The control group will receive an injection of 50mL of 0.9% sodium chloride solution.
  normal saline: Injection containing normal saline will be performed while the patient is still under general anesthesia, following wound closure, and will be injected evenly between the deep and superficial tissues in an extra-articular pattern (no injection of the synovium or capsule).
Period: Overall Study
Arm/Group | Pain Injection | Normal Saline
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Injection | Normal Saline | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (2.4) | 9.0 (2.9) | 8.6 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 12 | 8 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Average post-operative opioid consumption, measured in morphine equivalents per kilogram
Time Frame: During initial post-operative hospitalization (estimated 3-4 days)
Measure: Mean (Standard Deviation); unit: mEQ/kg
Arm/Group | Pain Injection | Normal Saline
Number analyzed (Participants) | 17 | 17
mEQ/kg | 0.41 (0.42) | 1.87 (2.05)

2. Secondary Outcome: Hospital Length of Stay
Description: Post-operative hospital length of stay
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pain Injection | Normal Saline
Number analyzed (Participants) | 17 | 17
days | 3.6 (2.3) | 3.4 (1.8)

3. Secondary Outcome: Post-operative Pain Scores
Description: Pain score assessments will be completed in the post-anesthesia care unit, & every 4 hours following surgical procedure. Scores will be collected by nursing staff on the inpatient ward who are blinded to treatment allocation and recorded in the electronic medical record. The type of pain score collection will vary based on patient age and level of intellectual disability. In verbal children, either the visual analog scale (VAS) or faces pain scale will be employed (scale 0-10; minimum 0, maximum 10). In non-verbal children, the Face, Legs, Activity, Cry, Consolability (FLACC) scale will be employed (scale 0-10; minimum 0, maximum 10). All 3 scales measure a patient's pain on a scale of zero (no pain) to ten (the worst pain). Lower values are considered better than higher values. These scores will be combined into an average score for the hospitalization. A higher average score indicates more pain (worse outcome), while a lower average score indicates less pain (better outcome).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pain Injection | Normal Saline
Number analyzed (Participants) | 17 | 17
scores on a scale | 1.0 (0.6) | 2.4 (1.1)

4. Secondary Outcome: Parent Satisfaction
Description: Parent satisfaction will be based on a standardized, validated questionnaire taken by parents in person at the first post-operative clinic visit aimed to assess their satisfaction with their child's pain management peri-operatively. Questions pertaining to pain interference are answered with a score of 1-5, with 1 being the best outcome and 5 being the worst outcome. Questions pertaining to severity of side effects are answered with a score of 0-10, with 0 being the best outcome and 10 being the worst outcome. Overall satisfiction is rated 1-5, with one being the best outcome and 5 being the worst. Finally, estimated time spent in severe pain is a percentage (0-100), with 0 being the best outcome and 100 being the worst. The score for each question are added to obtain a total score. A higher total score indicates a worse level of satisfaction with perioperative pain management. The scale goes from minimum 5 to maximum 155, with a score of 5 being the best and 155 being the worst.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Injection | Normal Saline
Number analyzed (Participants) | 12 | 15
score on a scale | 48.9 (30.6) | 47.3 (22.0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a minimum of 6 months postoperatively and a maximum of 3 years postoperatively.
Arm/Group | Pain Injection | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT04074265/Prot_SAP_001.pdf